CLINICAL TRIAL: NCT00829582
Title: Randomized, Placebo-Controlled, Double-Blind, Dose-Escalation Phase I Study of the Safety, Tolerability and Pharmacokinetics of a Single Intravenous Dose of ETI-204 (AnthimTM) [Elusys Protocol Number AH-102]
Brief Title: Intravenous Dose-Escalation Study With ETI-204 in Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elusys Therapeutics (Other)
Responsible Party: Irena Kirman, MD, PhD, Elusys Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AH-102
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2010-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — obiltoxaximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETI-204 (Experimental): ETI-204, Anthim
  Interventions: Drug: ETI-204, "Anthim"
- placebo (Sham Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: ETI-204, "Anthim" — single intravenous infusion of 120, 240 or 360 mg of ETI-204
  Arms: ETI-204
Other: placebo — single intravenous infusion
  Arms: placebo

SUMMARY:
Title: Randomized, Placebo-Controlled, Double-Blind, Dose-Escalation Phase I Study of the Safety, Tolerability and Pharmacokinetics of a Single Intravenous Dose of ETI-204 (AnthimTM)

Population: This study will determine the safety, tolerability and pharmacokinetics of a single iv dose of ETI-204 in subjects 18 to 50 years of age. Three cohorts will be studied sequentially: subjects receiving 120 mg, 240 mg and 360 mg of ETI-204. The study will be randomized, double-blind, and stratified by gender. Each cohort will contain 15 subjects (including at least four females), twelve who will receive ETI-204 and three who will receive placebo.

Study Objectives: To determine the safety, tolerability and pharmacokinetics of ETI-204 following a single intravenous administration.

DETAILED DESCRIPTION:
Study Duration: Maximum 70 days for each subject (from enrollment to end of follow-up period), unless the Day 70 HAHA (human anti-humanized antibodies) is positive, in which case subjects will be followed until HAHA test results are negative. This does not represent the total study duration, which is determined by the screening period and enrollment rate.

Description of Agent: ETI-204 is a monoclonal antibody (MAb) to protective antigen (PA) from Bacillus anthracis.

Schedule of Evaluations: Blood for pharmacokinetics (antibody concentration): Predose and at the following times after the start of infusion: 60 minutes (i.e., at the completion of the infusion), 3, 6, 12, 24 and 48 hours and on Days 7, 14, 21, 42, 56 and 70.

Blood chemistry, hematology, and urinalysis (referred to as safety laboratory assessments in the schedule of events), and urine drug screen (including ethanol and cotinine at all visits): Screening, Day 0, immediately pre-dose and on the following days after the start of infusion: 7, 14, 21, and 42. Urine pregnancy tests for all females will be performed at screening, baseline, immediately pre-dose and at 42 days. Tests of coagulation and viral serology tests will be done at screening only.

ECG: A 12-lead ECG will be done at screening. In subjects with acceptable ECG parameters, continuous 24-h Holter monitoring. will be then performed. After enrollment, a standard 12-lead ECG recording will be performed on study Day 1 (predose, 1.5h, 2h, 4h, 8h and 12h ±20 min) and continuous ECG telemetry monitoring beginning approximately 2 hours prior to the start of infusion and continuing at least 14 hours after the start of infusion. ECG is also recorded at the following study Days: 2, 7, 14, 21, and 42.

Measurement of product specific human anti-humanized antibodies (HAHA): Pre-dose and 42 days after dosing. HAHA positive subjects on Day 42 will be followed bi-weekly until study Day 70 and then monthly until HAHA test results are negative.

Vital signs (BP, P, T, RR): Screening, Day 0, before and at the following times after the start of the infusion on study day 1: 15, 30, 45, 60, 90±3 minutes; 2h,4h,8h, 12h and 24h±10 minutes (Day 2); Days 7, 14, 21 and 42.

Screening for Local and Systemic Adverse Events: The infusion site and proximal areas will be inspected for evidence of erythema, edema, visible or palpable cord, etc. on study days 1, 2, 7, 14, 21 and 42.

Participating Sites: The Ohio State University Clinical Pharmacology Unit Columbus, Ohio

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects between the ages of 18-50 inclusive at the time of enrollment. In each of the drug cohorts (subgroups), at least three of the subjects must be female.
2. The following screening laboratory parameters must be within 5% of the normal range: CBC (excluding WBC) and coagulation tests (aPTT, PT and INR). Absolute counts of WBC must be within 10% of the normal range. BUN, creatinine, and total and direct bilirubin may be up to 10% above the upper limits of normal. AST, ALT and alkaline phosphatase must be within normal limits. Urinalysis must be within generally accepted normal limits.
3. The values for the following tests at screening are to be:

   G-6-P dehydrogenase - normal HBsAg - negative HBV - negative (except immunized subjects may have positive anti-HBs) Anti-HCV - negative Anti-HIV (HIV antibody test) - negative Urine drug screen (including cotinine) - negative
4. Female subjects must agree to practice heterosexual abstinence or to use a licensed, effective form of birth control (e.g., oral contraceptives, diaphragm or condom in combination with contraceptive jelly, cream or foam, intrauterine contraceptive device, Depo-Provera®, skin patch, vaginal ring, or cervical cap) for at least 30 days prior to enrollment and for the duration of the study, including the follow-up period. Females using hormonal contraceptives must agree to use at least one other method for at least 30 days prior to enrollment and for the duration of the study, including the follow-up period.
5. Female subjects must have a negative pregnancy test.
6. No history of hospitalization for illness within the six months prior to study enrollment.
7. Nonsmoker or ex-smoker. If a subject is an ex-smoker, he/she must not have used nicotine for at least 6 months prior to enrollment. This will be confirmed by a negative urine test for cotinine. Exceptions may be made for sporadic users with negative urine cotinine tests; this will be determined on a case-by-case basis.
8. Able to spend the two days specified in the study schedule confined in a facility under study rules.
9. Able to read, understand and sign the informed consent form

Exclusion Criteria:

1. Routine consumption of any medication (prescription or OTC), vitamin, mineral, or dietary supplement, for one week before and during the study. The sole exceptions are hormonal contraceptive agents, as detailed above. The withdrawal time for any prescription medication should be no less than 1 week prior to the beginning of the study.
2. Blood pressure greater than 139 mm Hg systolic and 89 mm Hg diastolic. Repeat measurements are allowed.
3. Contraindication to the use of any monoclonal antibody: history of allergic reactions to any biologic or formulation component
4. Medical condition that in the Investigator's opinion could adversely impact the subject's participation, safety or conduct of the study.
5. Subject has taken an investigational medication in the previous three months.
6. The subject has a history of drug or alcohol abuse within the past two years.
7. The subject is female and plans to become pregnant during the whole study period or 6 months.
8. Calculated Body Mass Index (BMI) greater than 35.0 or less than 18.5.
9. The subject has been previously vaccinated with anthrax or has participated in clinical research involving anthrax.
10. Any ECG abnormality except for the following:

    * Sinus bradycardia, no lower than 46 beats per minute in younger, athletic subjects
    * Sinus tachycardia if the heart rate is within normal limits when vital signs are measured
    * Respiratory arrhythmia
    * Mild first degree A-V block (P-R interval < 0.23 sec)
    * Incomplete right bundle branch block
    * Left anterior hemiblock
    * Ectopic atrial focus
    * Premature atrial contractions
    * Unifocal premature ventricular contractions
    * Mild right or left axis deviation
    * Indeterminate axis
    * J-point elevation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Evidence of clinical safety following the infusion | 42 days

SECONDARY OUTCOMES:
immunogenicity | 42-70 days

CONTACTS AND LOCATIONS:
Overall Officials: Glen Apseloff, MD, Principal Investigator — OSU
Locations (1):
- Osu, 5084 Graves 333 W Tenth Ave, Columbus, Ohio, United States

REFERENCES:
- [Derived] Nagy CF, Leach TS, Hoffman JH, Czech A, Carpenter SE, Guttendorf R. Pharmacokinetics and Tolerability of Obiltoxaximab: A Report of 5 Healthy Volunteer Studies. Clin Ther. 2016 Sep;38(9):2083-2097.e7. doi: 10.1016/j.clinthera.2016.07.170. Epub 2016 Aug 24. PMID 27568215